CLINICAL TRIAL: NCT06505889
Title: Comparison of Low-cost Interventions for Pain Reduction During Radial Artery Puncture in the Emergency Department: A Three-arm Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 002/2567
Record Dates: First submitted 2024-07-01; First posted 2024-07-17 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Pain Control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three study groups (A, B, or C) to receive different local anesthesia methods prior to arterial blood sampling:
  Group A (Ice pack), Group B (10% lidocaine spray), Group C (Control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cryo-analgesic group (Ice pack) (Experimental): A standard cold pack chilled to -4°C will be applied to the arterial puncture site for 2 minutes. Following antiseptic cleaning and the physician will immediately perform the arterial blood sampling procedure with heparinized 3mL arterial blood gas syringe with a 22G x 1" needle.
  Interventions: Other: Local anesthesia methods
- Analgesic drug group (10% lidocaine spray) (Experimental): 10% lidocaine spray will be applied to the puncture site, covering a circular area (2-3 cm radius) around the puncture site for 2 minutes. Following antiseptic cleaning and the physician will immediately perform the arterial blood sampling procedure with heparinized 3mL arterial blood gas syringe with a 22G x 1" needle.
  Interventions: Other: Local anesthesia methods
- Control group (2% Chlorhexidine alcohol) (No Intervention): This group will receive standard antiseptic preparation with chlorhexidine in alcohol applied in a circular area (2-3 cm radius) around the puncture site for 2 minutes. Following antiseptic cleaning and the physician will immediately perform the arterial blood sampling procedure with heparinized 3mL arterial blood gas syringe with a 22G x 1" needle.

INTERVENTIONS:
Other: Local anesthesia methods — Local pain control method before arterial blood sampling procedure
  Arms: Analgesic drug group (10% lidocaine spray); Cryo-analgesic group (Ice pack)

SUMMARY:
The objective of this clinical trial is to investigate if local anesthesia using topical analgesic drug (10% lidocaine spray) or cryo-analgesic (Ice pack) can reduce pain levels during and after arterial blood sampling procedure. The research questions of this study includes:

* Can local anesthesia using topical analgesic drug (10% lidocaine spray) or cryo-analgesic (Ice pack) reduce pain levels during arterial blood sampling?
* Is the first-attempt success rate of arterial blood sampling higher when using local anesthesia (lidocaine spray or ice pack) compared to standard practice without anesthesia?

DETAILED DESCRIPTION:
This single center randomized controlled trial was conducted at the Emergency Department of Queen Savang Vadhana Memorial Hospital, Thailand.

Total of 126 Participants will be sequentially assigned to one of three study groups (A, B, or C) to receive different local anesthesia methods prior to arterial blood sampling procedure.

* Group A (Cold Application): A standard cold pack chilled to -4°C will be applied to the arterial puncture site for 2 minutes. Following cleaning, the physician will immediately perform the arterial blood sampling.
* Group B (Topical Anesthetic): 10% lidocaine spray will be applied to the puncture site, covering a circular area with a 2-3 cm radius. After allowing 2 minutes for anesthetic effect, the site will be cleaned and the physician will perform the arterial blood sampling.
* Group C (Control): This group will receive standard antiseptic preparation with chlorhexidine in alcohol applied in a circular area with a 2-3 cm around the puncture site. After 2 minutes, the site will be cleaned and the physician will perform the arterial blood sampling.

Participants will complete a questionnaire assessing pain levels both during and after the arterial blood sampling procedure. Arterial blood sampling procedure was conducted by trained research assistants or attending experienced physicians.

All collected data will be entered into a secure, encrypted form, ensuring patient confidentiality and preventing access to individual patient identifiers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, who present to the emergency department of Queen Savang Vadhana Memorial Hospital that requires arterial blood sampling procedure for diagnostic purposes

Exclusion Criteria:

* Altered level of consciousness (Glasgow Coma Scale < 15)
* Cognitive impairment or communication barriers precluding accurate pain assessment (e.g., severe dementia, aphasia, intoxication, delirium)
* Contraindications to radial artery cannulation (e.g., severe peripheral vascular disease, history of arteriovenous fistula at the puncture site, active infection at the puncture site)
* Pregnancy
* Need for emergency management which any delay could worsen patient care (e.g., cardiac arrest, respiratory failure requiring immediate intubation)
* Known allergy or hypersensitivity to lidocaine or amide-type local anesthetics
* Severe pain from other sources that could distracting pain assessment related to the arterial blood sampling procedure (e.g., significant trauma, bone fractures, severe burns)
* Failure to obtain successful arterial access after two attempts by an experienced operator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Pain score both during and after the arterial blood sampling procedure. | Participants will rate their pain score both during and at 30 seconds after the arterial blood sampling procedure.
  Pain score will be assessed using a horizontal numeric Rating Scale (NRS) ranging from 0 to 10, with 0 representing "no pain" and 10 representing "the worst pain."

SECONDARY OUTCOMES:
The first-attempt success rate for arterial blood sampling procedure when using local anesthesia. | During the arterial blood sampling procedure.
  First-attempt success refer to blood sample being successfully drawn from the radial artery at the first trial of skin penetration without needle being withdrawn
explore the relationship between associated factors and overall time for arterial blood draw. | procedure time was recorded since intervention was performed by physician. end point is when physician withdraw an ABG needle from patient skin.
  Multivariate linear regression analysis was performed to determine factors associated with time taken for arterial blood draw.

CONTACTS AND LOCATIONS:
Overall Officials: Chawin Taveekijakarn, MD, Principal Investigator — QSMVH
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Chon Buri, Thailand